CLINICAL TRIAL: NCT06757361
Title: Effect of Screen Time Exposure on Eating Behaviour and Health Related Quality of Life in Normal Preschool Children
Brief Title: Effect of Screen Time Exposure on Eating Behaviour and Health Related Quality of Life
Status: Active, not recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mennatallah Galal Mohamed Hassanein, Principal investigator, Cairo University
Other Study IDs: P.T.REC/012/005461
Record Dates: First submitted 2024-12-12; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Eating Behavior Disorders; Health-Related Quality of Life; Screen Time Exposure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to learn the effect of screen time exposure on eating behaviour and health related quality of life in normal preschool children.

DETAILED DESCRIPTION:
Screen media devices have become an integral to daily life, especially for preschool children due to emerging technologies, increased marketing , widespread familial and societal use , and easy access to or ownership for young children. Common screen activities include watching television, digital video discs and videos, playing video games, and using apps . However ,excessive screen time, non-educational screen content, unsupervised and early screen exposure can have numerous potential negative effects on children's health .

Screen time can significantly affect quality of life in various ways, both positively and negatively. Regarding cognitive development, screens have the potential to enhance education and learning. However, studies have shown that excessive screen time can negatively affect executive functioning, sensorimotor development, and academic outcomes. Early screen exposure has been associated with lower cognitive abilities and academic performance in later years. Language development is also affected by screen time, as it diminishes the quantity and quality of interactions between children and caregivers. Excessive screen usage can also lead to problems in social-emotional development, including obesity, sleep disturbances, depression, and anxiety. It can impair emotional comprehension, promote aggressive behavior, and hinder social and emotional competence .

ELIGIBILITY:
Inclusion Criteria

1. Chronological age range 5 :6
2. Both genders will be included
3. According to score of screen dependency scale children stratified into Two Groups:

   * Group A children score more than 24.5
   * Group B children score less than 24.5

Exclusion Criteria:Any children has one or more from the following criteria:

1. Any surgical intervention in mouth.
2. Any congenital anomaly in the mouth as cleft lips or cleft palate.
3. Oral disorders

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 1. Chronological age range 5 :6
  2. Both genders will be included
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Eating Behavior in Preschool Children | 12 weeks
  Eating behaviour will be assessed in preschool children using a validated tool that evaluates overall eating habits, including Food Responsiveness, Enjoyment of Food, Emotional Overeating, Desire to Drink, Satiety Responsiveness, Slowness in Eating, Emotional Undereating, and Food Fussiness.
Health-related quality of life (HRQoL) | 12 weeks
  Health-related quality of life (HRQoL) will be assessed in preschool children using a validated measurement tool. This tool evaluates the child's overall well-being, considering physical, emotional, social, and school functioning as part of a comprehensive assessment of quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy Cairo university, Helwan, Helwan, Egypt

IPD SHARING:
Plan to Share IPD: No